CLINICAL TRIAL: NCT03431844
Title: Prospective Clinical Observational Study of Humanin Isoforms in Cardiac Muscle and Blood Plasma and Their Association to Major Complications After Cardiac Operation
Brief Title: Humanin Isoforms in Cardiac Muscle and Blood Plasma and Major Complications After Cardiac Operation
Status: Completed | Type: Observational
Sponsor: University of Tartu (Other)
Collaborators: Tartu University Hospital (Other); North Estonia Medical Centre (Other)
Responsible Party: Principal Investigator, Henery Kroon, Researcher, University of Tartu
Other Study IDs: HN1160
Record Dates: First submitted 2018-01-18; First posted 2018-02-13 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Myocardial Ischemia; Coronary Artery Bypass Surgery
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Right atrial heartmuscle biopsy, blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective of the study is to clarify humanin-like peptide concentration in myocard tissue and in blood and to study if its concentration level is related to early complication occurrence and frequency after cardiac operation.

Hypothesis of the study is that previously described elements are related to each other.

DETAILED DESCRIPTION:
Data collection: Historical medical and preoperative data, operation data (type of operation performed and its details), detailed postoperative course (occurrence of complications).

Specimen collection:

* Tissue sample is taken during the operation from the right atrial appendage of the heart and the sample is frozen at -80 C.
* Blood samples are taken just before the operation, one hour after aortic cross-clamp removal and the next morning after the operation. Samples are processed and blood plasma is frozen at -80 C.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years
* Ischemic heart disease in medical history
* Planned on-pump coronary artery bypass graft (CABG) operation
* Signed informed consent by patient

Exclusion Criteria:

* Age <18 years
* Planned isolate valve or aortic operation
* Patient is in another study with an intervention
* Absence of signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients who have a history of ischemic heart disease and who are going to have an elective on-pump CABG operation.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days
  30-day all-cause mortality
Major complications: myocardial infarction. | 30 days
  Diagnosed myocardial infarction.
Major complications: acute kidney injury. | 30 days
  Diagnosed acute kidney failure (KDIGO stage).
Major complications: stroke. | 30 days
  Diagnosed stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Starkopf, MD, PhD, Study Director — Tartu University Hospital
Locations (2):
- Estonia (2):
  - North Estonia Medical Centre, Tallinn, Harju
  - Tartu University Hospital, Tartu, Tartu